CLINICAL TRIAL: NCT03173183
Title: Clinical Research on Treatment of Functional Dyspepsia With Genuine Regional Rhizoma Atractylodis: a Randomized Double-blind Placebo Controlled Trial
Brief Title: Treatment of Functional Dyspepsia With Genuine Regional Rhizoma Atractylodis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yanming Xie, Executive director, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2060302-1401-03
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Efficiency of Genuine Regional and Non-genuine Regional Rhizoma Atractylodis in Treating FD

STUDY DESIGN:
Intervention Model Description: The research is designed by randomized, double-blind, placebo and parallel clinical control.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- genuine regional Rhizoma Atractylodis (Experimental): Granules of genuine regional Rhizoma Atractylodis:
  Maozhu granule, 9g per bag, manufactured by Guangdong Yifang Pharmaceutical Co., Ltd., orally administration, 9g per time, 3 times a day.
  Interventions: Drug: genuine regional Rhizoma Atractylodis (Maozhu granule)
- non-genuine regional Rhizoma Atractylodis (Active Comparator): Granules of non-genuine regional Rhizoma Atractylodis (Luotian, Hubei province) :
  Luozhu granule, 9g per bag, manufactured by Guangdong Yifang Pharmaceutical Co., Ltd., orally administration, 9g per time, 3 times a day.
  Interventions: Drug: genuine regional Rhizoma Atractylodis (Maozhu granule)
- placebo (Placebo Comparator): placebo granules: Simulants (granule), 9g per bag, manufactured by Guangdong Yifang Pharmaceutical Group Co., Ltd., orally administration, 9g per time, 3 times a day.
  Interventions: Drug: genuine regional Rhizoma Atractylodis (Maozhu granule)

INTERVENTIONS:
Drug: genuine regional Rhizoma Atractylodis (Maozhu granule) — Maozhu granule, 9g per bag, manufactured by Guangdong Yifang Pharmaceutical Co., Ltd.
  Luozhu granule, 9g per bag, manufactured by Guangdong Yifang Pharmaceutical Co., Ltd.
  Simulants (granule), 9g per bag, manufactured by Guangdong Yifang Pharmaceutical Group Co., Ltd.
  Other Names: non-genuine regional Rhizoma Atractylodis (Luozhu granule); placebo granules

SUMMARY:
This is a randomized double-blind placebo controlled trial aim to compare the efficiency of genuine regional and non-genuine regional Rhizoma Atractylodis in treating functional dyspepsia. This study will also observe the clinical safety of genuine regional Rhizoma Atractylodis.The trial will be conducted in Xiyuan Hospital of China Academy of Chinese Medicine Sciences and Dongzhimen Hospital of Beijing University of Chinese Medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the FD Rome Ⅲ diagnosis standard;
2. Meeting TCM differentiated diagnosis standard of the spleen deficiency with dampness pattern;
3. Without taking any medicines affecting gastric motility in the recent 14 days;
4. Between 18 and 65 years old;
5. Voluntary participation in the trial and signing informed consent.

Exclusion Criteria:

1. Combined irritable bowel syndromes; combined peptic ulcer, erosive gastritis, atrophic gastritis, abdominal surgery history, gastric mucosa with severe dysplasia or pathological diagnosis of suspected malignant transformation; combined gastroesophageal reflux disease, irritable bowel syndrome with overlapping syndromes.
2. Patient whose differentiation is not clear or who doesn't belong to the spleen deficiency with dampness pattern.
3. Women in pregnancy, breastfeeding or have fertility plans recently; the legally disabled (blind, deaf, dumb, mental retardation, mental disorders, physical disability)
4. Patients with endocrine and metabolic diseases such as connective tissue diseases, diabetes, menopausal syndromes; patients combined with heart rate disorder, severe diseases in cardiovascular, brain, liver, lung, kidney and hematopoietic systems, acute and chronic infectious diseases, malignant tumors, mental illness.
5. Allergy to the trial drug.
6. With suspected or definite alcohol, drug abuse history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
disappearance rate of dyspepsia | Eight weeks
  The evaluation is divided into five levels: symptoms disappeared; significant improved; moderate improved, no change; deteriorated.

SECONDARY OUTCOMES:
The Short-Form Leeds Dyspepsia Questionnaire, SF-LDQ | Eight weeks
Nepean Dyspepsia Index, NDI | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, M.D., Principal Investigator — China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No